CLINICAL TRIAL: NCT01271426
Title: Association of Complement Factor H and ARMS2 Genotypes With Response of Polypoidal Choroidal Vasculopathy to Intravitreal Ranibizumab
Brief Title: Response to Ranibizumab in Polypoidal Choroidal Vasculopathy (PCV)and SNPs
Status: Completed | Type: Observational
Sponsor: Nihon University (Other)
Other Study IDs: NihonU-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal Choroidal Vasculopathy; Ranibizumab
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — white blood cell

SUMMARY:
To determine whether complement factor H (CFH) and age-related maculopathy susceptibility 2 (ARMS2) genotypes have a pharmacogenetic effect on the treatment of polypoidal choroidal vasculopathy (PCV) with ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Polypoidal choroidal vasculopathy
* must have injection of Ranibizumab

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients in hospital
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Association of Complement Factor H and ARMS2 Genotypes with Response of Polypoidal Choroidal Vasuculopathy to Intravitral Ranibizumab | a month after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Surugadai Nihon university hospital, 1-8-13 Kandasurugadai Chiyoda-ku, Tokyo, Japan